CLINICAL TRIAL: NCT05917847
Title: Awake VDL Intubation With Dexmedetomidine, a Case Series
Brief Title: Awake VDL Intubation With Dexmedetomidine, a Case Series (DexAwake)
Acronym: DexAwake
Status: Completed | Type: Observational
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Elena Cagnazzi, DM, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: DA001
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Awake Intubation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Awake intubation — Awake videolaryngoscopic intubation with dexmedetomidine for sedation

SUMMARY:
Early after the videolaryngoscope'(VDL) introduction in clinical practice, the awake videolaryngoscopic (A-VDL) intubation took place with and instead of the awake video-bronchoscopic (A- VBS) intubation. The awake intubation is a safe profile technique that was underused since the only instrumentation available was the fiberoptic bronchoscope (FOB) or more recently the video-bronchoscope (VBS). With the VDL diffusion, the awake intubation option has eventually turned into a more utilized procedure, with the potential to become a daily procedure. This was also due to dexmedetomidine (DEX) introduction in The Operating Room pharmacopeia. Several steps must be standardized in order to homogeneously apply an awake intubation protocol. A department protocol is recommended (awake intubation guidelines) but a low threshold for enrollment can be used to shorten and standardize the execution times. This study aims to create a protocol and measure the outcomes.

DETAILED DESCRIPTION:
Early after the videolaryngoscope'(VDL) introduction in clinical practice, the awake videolaryngoscopic (A-VDL) intubation took place with and instead of the awake video-bronchoscopic (A- VBS) intubation. The awake intubation is a safe profile technique that was underused since the only instrumentation available was the fiberoptic bronchoscope (FOB) or more recently the video-bronchoscope (VBS). With the VDL diffusion, the awake intubation option has eventually turned into a more utilized procedure, with the potential to become a daily procedure. This was also due to dexmedetomidine (DEX) introduction in The Operating Room pharmacopeia.

The emergency use of rescue techniques after failed intubation throws the operator into the rare, but unwanted emergency "Front of Neck Access" (FONA) scenario, while a failed awake intubation brings (carry, get) the operator into the "patient not intubated but safely and spontaneously breathing" scenario, moving away from the events of hypoxic complications and death.

Several steps must be standardized in order to homogeneously apply an awake intubation protocol. First, the patients need to be clinically evaluated for difficult intubation predictors. Most of the articles about prediction only investigated the relationship between difficult intubation' predictors and direct laryngoscopy and they showed poor to moderate sensitivity and specificity (Toshiga Shiga, Vannucci) but, moving on VDL' world this relationship has changed as showed by Cortellazzi et al with an AUC for El Ganzouri Risk Index improving from 0.74 to 0.9 using DL and Glidescope respectively. In addition to these considerations, all the most recent Airway Management Guidelines has confirmed as unmissable the clinical evaluation of anthropometric and clinical DI predictors. (DAS) Along with measuring all the EGRI parameters, it is pivotal to examine any abnormality in the head, pharyngo-laryngeal, neck, spine, and abdominal anatomy. Previous neck irradiation, mass lesions, neck circumference, super-obesity, severe cervico-dorsal kyphosis, or past pharyngo-laryngeal surgery have to be considered and may not alter the EGRI score that is, incidentally, made -as the other predictors -for apparently normal patients (Shiga).

A department protocol is recommended (awake intubation guidelines) but a low threshold for enrollment can be used to shorten and standardize the execution times.

We retrospectively evaluated 24 patients (from January 2019 to June 2021). For descriptive purposes, there are five procedural "Times": T0, T1, T2, T3, T4 and T5. T 0 is the start of the dexmedetomidine charge dose and local oral-pharyngeal anesthetic. In T1, the GAG reflex check is performed. In T2 fentanyl or ketamine is delivered. In T3 the local anesthetic is nebulized on vocal cord and trachea, under videolaryngoscopic view. T4 is the tube passage through the vocal cords. T5 is the EtCo2 curve assessment. At the end outcomes were measured.

ELIGIBILITY:
Inclusion Criteria:

* Abnormality in the head, pharyngo-laryngeal, neck, spinal anatomy, super-obesity, El Ganzouri Risk Index > 6 or high risk for ab ingestis or hemorrhage (i.e.: tongue, pharynx-hypopharynx cancer lesions or arteriovenous malformations)

Exclusion Criteria:

* Interdental distance <1 cm
* Need for emergency airway stabilization.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
The number of A-VDL success | from the starting of sedation to the end of the intubation procedure
  This was defined as the ability to identify good or poor glottic view without rupture of sedation or change in Rass/Ramsay sedation level.
The number of A-VDL intubation successes | from the starting of sedation to the end of the intubation procedure
  This was defined as the number of effective tube passages and airway stabilization.

SECONDARY OUTCOMES:
Number of intubations allocated after A-VDL to VBS intubation. | from the starting of sedation to the end of the intubation procedure
  Airway stabilization
The kind of drugs used and dosage | from the starting of sedation to the end of the intubation procedure
  Type of drug and dosage
Level of sedation obtained | from the starting of sedation to the end of the intubation procedure
  Rass/ Ramsay
Presence absence of memory of pain or discomfort during the procedure | from the starting of sedation to the end of the intubation procedure
  Pain or discomfort remembered by the patient
Presence/absence of complications | from the starting of sedation to the end of the intubation procedure
  procedure abandonment for reasons other than poor glottic visualization, desaturation above 90%, bradycardia above 40

OTHER OUTCOMES:
Minutes from the beginning of sedation until airway stabilization | from the starting of sedation to the end of the intubation procedure
  Time in minutes
Cormack and Lehane score obtained | from the starting of sedation to the end of the intubation procedure
  C&L

CONTACTS AND LOCATIONS:
Overall Officials: Elena Cagnazzi, MD, Principal Investigator — Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Locations (1):
- Spedali Civili, Brescia, Italy